CLINICAL TRIAL: NCT02857465
Title: Epidural Dexamethasone for Labor Analgesia: the Effects on Ropivacaine Consumption and Labour Outcome. A Randomized Double Blind Placebo Study
Brief Title: Epidural Dexamethasone for Labor Analgesia: the Effects on Ropivacaine Consumption and Labour Outcome
Acronym: DEXAPER
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: French Agency for the Safety of Health Products refusal
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/CHU/12
Record Dates: First submitted 2016-07-26; First posted 2016-08-05 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Obstetric Pain; Other Complications of Obstetric Anesthesia - Delivered
MeSH Terms: conditions — Labor Pain | interventions — Dexamethasone; Ropivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural analgesia + DEXAMETHASONE (Experimental): Single epidural injection of Dexamethasone Mylan (8 mg) concomitant to epidural analgesia (ropivacaine+ sufentanil)
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine; Drug: Sufentanil
- Epidural analgesia + PLACEBO (Placebo Comparator): Single epidural injection of sodium chloride (0.9%) Lavoisier concomitant to epidural analgesia (ropivacaine + sufentanil)
  Interventions: Drug: Placebo; Drug: Ropivacaine; Drug: Sufentanil

INTERVENTIONS:
Drug: Dexamethasone — single epidural injection of dexamethasone (8 mg) in addition to local anesthetics used for epidural analgesia
  Other Names: Dexamethasone MYLAN
  Arms: Epidural analgesia + DEXAMETHASONE
Drug: Placebo — single epidural injection of sodium chloride 0.9% (2 mL) in addition to local anesthetics used for epidural analgesia
  Other Names: Sodium chloride LAVOISIER 0.9 %
  Arms: Epidural analgesia + PLACEBO
Drug: Ropivacaine — NAROPEINE 7.5 mg/mL is diluted at the concentration of 1 mg/mL prior to the epidural use. The perfused dose depends on the efficacy of analgesia in reducing the delivery labor pain.
  Other Names: NAROPEINE 7.5 mg/ml; anhydrous ropivacaine chlorhydrate
Drug: Sufentanil — Sufentanil 0.5 mg/L is used as solution for injection for epidural analgesia and used in combination with ropivacaine. The administered dose is bolus of 15 to 20 micrograms diluted into 10 mL.
  Other Names: Sufentanil Mylan 0.5 microg/mL

SUMMARY:
To assess the efficacy of epidural dexamethasone administration, compared to placebo, in reducing local anesthetics consumption during labor epidural analgesia in parturient women

DETAILED DESCRIPTION:
It is hypothesized that reducing the consumption of local anesthetics during labor epidural analgesia could lower their side effects (rate of motor block, nausea and emesis during labor, maternal hypotension, maternal fever) and improve the duration of the second part of the labor, and the new-born adaptation to child-birth and during the first 24 hours. The use of instruments for assisted vaginal delivery and the needs to perform emergency cesarean could also be impacted.

The efficacy of the dexamethasone will be assessed by the hourly Ropivacaine consumption (milligrams/hour) measured from randomization time to the end of epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* First and single pregnancy, Full term (> 37 wks amenorrhea), Cephalic presentation, Spontaneous labor, Epidural analgesia requested by the parturient

Exclusion Criteria:

* Minor patient, Planned cesarean section, Gestational hypertension and preeclampsia, Gestational diabetes, opioids or ocytocin administration before epidural analgesia preparation, Allergy to dexamethasone, Untreated gastroduodenal ulcer, epidural analgesia contraindications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Hourly ropivacaine consumption expressed as mg/mL used during epidural analgesia in parturient women | From the beginning to the end of epidural analgesia, that could last up to 6 hours
  The administered dose of ropivacaine during epidural is used to measure the efficacy of Dexamethasone in reducing local anesthetics during labor analgesia

SECONDARY OUTCOMES:
Improvement of epidural analgesia assessed by the reduction of adverse effects induced by local anesthetics | From the beginning to the end of epidural analgesia, that could last up to 6 hours
  Adverse effects such as nausea and emesis, maternal hypotension, maternal hyperthermia will be recorded during epidural analgesia
Dexamethasone effect maternal pain during delivery assessed by Visual Analogic Scale | From the beginning to the end of epidural analgesia, that could last up to 6 hours
  Evaluation of the lowered maternal pain induced by Dexamethasone
Improvement of delivery assessed by recording the number of side events (motor block, emergency cesarean, instrument-assisted delivery) | From the beginning to the end of epidural analgesia, that could last up to 6 hours
  Rates of motor block, emergency cesarean, instrument-assisted delivery
Maternal satisfaction assessed by visual analogic scale | On the morning of the next day after delivery, up to 24 hours
  Patient satisfaction visual analogic scale

OTHER OUTCOMES:
New-born adaptation to child-birth assessed by "Apgar score" | up to 5 minutes after child-birth
  Apgar score assessed twice: at 1 minute and 5 minutes after child-birth
New-born adaptation to child-birth assessed by umbilical biochemical parameters | umbilical blood collection up to 5 minutes after child-birth
  Measurement of umbilical pH and lactates values at child-birth
New-born adaptation to child-birth assessed by the rate of neonatal respiratory distress | 0-24 hours after child-birth
  Rate of neonatal respiratory distress during the first 24 hours after child-birth

IPD SHARING:
Plan to Share IPD: No